CLINICAL TRIAL: NCT06916845
Title: Data Collection for CapsoView AI Software Development for the CapsoCam® Colon (CV-3E)
Brief Title: Data Collection for CV-3E AI Software Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capso Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLN-CVI-7472
Record Dates: First submitted 2025-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Participants (Experimental): All participants will swallow the CapsoCam® Colon (CV-3E).
  Interventions: Device: Colon Capsule

INTERVENTIONS:
Device: Colon Capsule — All participants will swallow the CapsoCam® Colon (CV-3E) for this study.

SUMMARY:
The goal of this clinical trial is to collect capsule images for the development of CADe software for use with the CapsoCam® Colon (CV-3E) in healthy volunteers who have been referred for colonoscopy. There will be no analysis performed as part of this protocol.

Participants will

* adhere to bowel prep instructions and dietary requirements
* ingest pro-kinetic medication and CapsoCam® Colon (CV-3E)
* adhere to booster regimen and dietary requirements until capsule passes
* retrieve capsule with retrieval kit per instructions and mail back to sponsor
* participate in follow-up phone call

ELIGIBILITY:
Inclusion Criteria:

1. 45-75 years of age
2. Choose to participate and must have signed the IRB-approved informed consent document.

Exclusion Criteria:

1. Colonoscopy or CT-colonography within the past 5 years that demonstrated no polyps
2. Colonoscopy within the past 4 years that demonstrated polyps that were removed.
3. Has contraindication for capsule endoscopy
4. Subject is suspected or diagnosed with familial adenomatous polyposis, hereditary non polyposis colon cancer, or any high-risk genetic syndrome
5. Subject is suspected or diagnosed with inflammatory bowel disease such as ulcerative colitis or Crohn's disease
6. History of incomplete colonoscopy
7. Type I or uncontrolled II Diabetes (Uncontrolled defined as HbA1C>6.4 within the past 3 months and/or with history of constipation or gastroparesis).
8. Impaired cardiac function assessed as greater than NYHA Class II
9. History of small- or large-bowel obstructive condition
10. Known history of swallowing disorder, and/or ischemic bowel disease neuropathies and/or radiation enteritis
11. Known history of NSAID enteropathy and stricture resulting from taking NSAIDs on a regular basis that, in the opinion of the Investigator, would put the subject at greater risk for capsule endoscope retention
12. Known allergy to ingredients used in bowel preparation and boosters
13. Daily and/or regular narcotic use
14. Decompensated cirrhosis
15. Prior abdominal radiation therapy
16. Diagnosis of anorexia or bulimia
17. History of or suspicion of any of the following: strictures, volvulus or intestinal obstruction, or internal hernias or abdominal surgeries that the Investigator believes should exclude the patient from study participation
18. Known or suspected megacolon
19. Scheduled to undergo MRI examination within 7 days after ingestion of the capsule
20. Has known slow gastric-emptying time or confirmed diagnosis of gastroparesis
21. Pregnant or nursing or of child-bearing potential and does not agree to practice medically acceptable methods of contraception. Women of child bearing potential (WOCBP) must have a negative urine pregnancy test at screening.
22. Unable to follow or tolerate fasting, bowel preparation, and other study procedures
23. Any documented medical or psychological condition or significant concurrent illness which, in the Investigator's opinion, would make it unsafe for the subject to participate in this research study or would affect the validity of the study results
24. Are currently enrolled in an interventional clinical study or currently enrolled in or within the last 30 days, a pharmaceutical clinical study
25. Chronic constipation as defined by <3 bowel movements per week, or the use of routine laxatives (other than fiber) to attain regular bowel movements

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Collect Capsule Images | 4-6 months
  No assessment will be done for this protocol. Videos will be collected for AI development for use in future study.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Digestive Diseases Center of Hattiesburg, LLC, Hattiesburg, Mississippi
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No